CLINICAL TRIAL: NCT04022499
Title: Enhanced Enrollment in the National Diabetes Prevention Program for the Underserved: a Randomized Control Trial
Brief Title: Presessions for the National Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-2542
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-05

CONDITIONS: Prediabetic State; Obesity; Gestational Diabetes
MeSH Terms: conditions — Prediabetic State; Obesity; Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-NDPP (Experimental): Presessions + usual care NDPP
  Interventions: Behavioral: Presessions; Behavioral: National Diabetes Prevention Program
- Usual care NDPP (Active Comparator): Usual care NDPP only
  Interventions: Behavioral: National Diabetes Prevention Program

INTERVENTIONS:
Behavioral: Presessions — The Pre-NDPP arm includes a "pre-session" with three components: 1) education about diabetes risks, 2) motivational interviewing (MI) to encourage participation in the NDPP and, 3) problem-solving of barriers to engagement.
  Arms: Pre-NDPP
Behavioral: National Diabetes Prevention Program — The Diabetes Prevention Program was a successful clinical trial demonstrating that intensive lifestyle support for weight loss reduced diabetes incidence by 58%. The intervention was translated into the National Diabetes Prevention Program (NDPP) and disseminated by the Centers for Disease Control and Prevention as a yearlong group-based program since 2012.

SUMMARY:
The National Diabetes Prevention Program (NDPP) is a widely available, evidence-based intervention that promotes weight loss to prevent type 2 diabetes; however, participant attendance is problematic and leads to suboptimal weight loss, especially among Hispanic, non-Hispanic black, and low-income non-Hispanic white participants. An innovative pre-session enhancement to the NDPP (Pre-NDPP) showed successful results upon initial application in a diverse and predominately low-income population, with doubled attendance and weight loss outcomes as compared to previous NDPP participants who did not receive a pre-session. If Pre-NDPP is shown to be successful upon more rigorous study, it can be widely adopted by NDPP providers across the country to help reduce diabetes prevalence and related health disparities.

DETAILED DESCRIPTION:
Type 2 diabetes affects 9.4% of US adults with higher rates among racial/ethnic minorities and individuals of low socioeconomic status. The National Diabetes Prevention Program (NDPP) is an evidence-based and widely disseminated behavioral intervention to reduce diabetes incidence through modest weight loss. However, retention in the yearlong NDPP is problematic and leads to suboptimal weight loss, especially among Hispanic, non-Hispanic black, and low-income non-Hispanic white participants. Strategies to improve NDPP engagement and weight loss are needed urgently, especially for these subgroups. Pilot results of the Pre-NDPP, a novel enhancement to enrollment in the NDPP based on the Health Belief Model, were highly successful in a non-randomized cohort study among 1,140 racially diverse, predominately low-income participants. Outcomes of 75 Pre-NDPP participants who enrolled in the NDPP were compared to 1,065 prior participants using ANCOVA and multivariable logistic regression. Pre-session participants stayed in the NDPP 99.8 days longer (p<.001) and attended 14.3% more sessions (p<.001) on average than those without a pre-session. Pre-session participants lost 2.0% more weight (p<.001) and were 3.5 times more likely to achieve the 5% weight loss target (p<.001). Sensitivity analyses were consistent. Findings suggest pre-sessions may be a promising and pragmatic strategy to improve NDPP effectiveness and mitigate disparities in program outcomes, but a randomized controlled trial (RCT) is needed to determine whether Pre-NDPP reliably improves NDPP outcomes. The purpose of this study is to 1) conduct an RCT comparing NDPP attendance and weight loss outcomes between participants who receive Pre-NDPP vs. direct enrollment into the NDPP (usual care), 2) examine potential effect mediators (perceived risk for developing diabetes and self-efficacy and readiness for weight control) and moderators (race/ethnicity and income level), and 3) evaluate implementation factors, including cost and projected return on investment. The long-term goal is to disseminate a scalable, evidence-based strategy to improve success of the NDPP and reduce disparities in NDPP effectiveness. If found to be effective, Pre-NDPP can be disseminated to all NDPP providers, including more than 1,700 NDPP sites, and may be supported by current NDPP payers such as Medicare, commercial insurers, and employer groups. Thus, this approach has a high potential to impact the burden of type 2 diabetes and related health disparities across the country.

ELIGIBILITY:
Inclusion Criteria:

* Denver Health patients
* BMI≥25 (≥23 if Asian)
* History of recent prediabetes or former gestational diabetes (GDM) diagnosis (patients without known prediabetes or past GDM may also be eligible based on a risk screening tool)

Exclusion Criteria:

* Pregnant at enrollment
* Known to have diabetes
* Non-English or non-Spanish-speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 483 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ritchie ND, Holtrop JS, Gritz RM, Sauder KA, Durfee MJ, Dickinson LM, Kaufmann PG. Enhanced Enrollment in the National Diabetes Prevention Program to Increase Engagement and Weight Loss for the Underserved: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Jun 1;9(6):e15499. doi: 10.2196/15499. PMID 32476659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We will identify potential participants through referrals from Denver Health healthcare providers to the Denver Health NDPP, per routine practice since 2013. Providers refer through the electronic health record (EHR), following email prompts to provider listservs in the preceding months of a new NDPP starting. Recruitment efforts began summer 2019 and concluded winter 2023.
Period: Overall Study
Arm/Group | Pre-NDPP | Usual Care NDPP
Started | 244 | 239
Completed | 236 | 234
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-NDPP | Usual Care NDPP | Total
Number analyzed (Participants) | 244 | 239 | 483
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (13) | 47.0 (12.9) | 46.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 190 | 382
  Male | 52 | 49 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: Percent body weight change from baseline to 12 months
Time Frame: 12 months
Population: Patients that were pregnant were excluded from the analysis
Measure: Mean (Standard Deviation); unit: % of weight loss
Arm/Group | Pre-NDPP | Usual Care NDPP
Number analyzed (Participants) | 236 | 234
% of weight loss | 3.1 (6.7) | 2.8 (6.0)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Description: Adverse events were not collected
Arm/Group | Pre-NDPP | Usual Care NDPP
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
A primary limitation of the randomized controlled trial (RCT) is that the planned sample size was calculated based on effect size data from an in-person NDPP pilot study, however, due to the Coronavirus Disease 2019 (COVID-19) pandemic, the RCT intervention was conducted as a virtual program. A smaller effect size for the virtual program may have resulted in the study being underpowered to detect a statistical difference between the two groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT04022499/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT04022499/ICF_001.pdf